CLINICAL TRIAL: NCT07185711
Title: Tooth Stability Assessment in Cemento-Osseous Dysplasia Using Resonance Frequency Analysis and Bite Force Sensor
Brief Title: RFA and Bite Force in COD Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Ömür Dereci, Prof., Eskisehir Osmangazi University
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EskisehirOU-Dereci-001
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Tooth Ankylosis; Cemento-Osseous Dysplasia; Jaw Diseases / Diagnosis
Keywords: pathology; Resonance Frequency Analysis; Bite Force
MeSH Terms: conditions — Tooth Ankylosis; Cementoma; Jaw Diseases; Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Teeth with Cemento-Osseous Dysplasia (Experimental): Teeth associated with cemento-osseous dysplasia were evaluated using Resonance Frequency Analysis (RFA) and a bite force sensor to assess ankylosis and stability.
  Interventions: Diagnostic Test: Resonance Frequency Analysis (RFA); Diagnostic Test: Bite Force Sensor
- Arm 2: Healthy Contralateral Teeth (Control Group) (Active Comparator): Healthy contralateral teeth from the same patients, without cemento-osseous dysplasia, were evaluated using the same methods (RFA and bite force sensor) for comparison with COD-associated teeth.
  Interventions: Diagnostic Test: Resonance Frequency Analysis (RFA); Diagnostic Test: Bite Force Sensor

INTERVENTIONS:
Diagnostic Test: Resonance Frequency Analysis (RFA) — Resonance frequency analysis performed with the Osstell™ device. SmartPeg was attached with composite resin to the occlusal surface of the tooth, and ISQ values were recorded in mesio-distal and bucco-lingual directions.
Diagnostic Test: Bite Force Sensor — Assessment of maximum bite force using a bite force sensor. Measurements were performed on COD-associated teeth and contralateral healthy controls for comparison.

SUMMARY:
This study aims to evaluate the periodontal attachment and ankylosis status of teeth associated with cemento-osseous dysplasia (COD). Using resonance frequency analysis (RFA) and a bite force sensor, the stability of COD-associated teeth was measured and compared with contralateral healthy teeth. These non-invasive and objective methods are expected to reveal the impact of COD lesions on the surrounding dentoalveolar structures.

DETAILED DESCRIPTION:
Cemento-osseous dysplasias represent the most common group of benign fibro-osseous lesions, frequently detected in the mandible and often asymptomatic. Although they generally do not require treatment, the remodeling of bone and cementum-like tissues around the tooth roots has clinical significance in terms of periodontal attachment and ankylosis. The present study aims to investigate the ankylosis status of teeth associated with COD lesions at different stages by using objective measurement tools.

In each patient, COD-associated teeth and contralateral healthy teeth were evaluated. Measurements were performed using resonance frequency analysis (RFA) with the Osstell™ device and additionally by a bite force sensor to assess functional stability. For RFA, SmartPeg magnetic attachments were fixed to the occlusal surface with composite resin, and three measurements were obtained in both mesio-distal and bucco-lingual directions. Mean ISQ values were then recorded. After measurements, SmartPeg was carefully removed without leaving residues, and patient comfort was evaluated using a six-point numeric rating scale.

The obtained RFA and bite force values will be statistically analyzed to compare COD-associated teeth with healthy controls. Furthermore, the study seeks to determine differences in ankylosis tendency across various COD stages and their potential impact on periodontal ligament integrity. This approach may provide valuable insights for understanding the clinical course of COD and for planning surgical interventions in symptomatic cases

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cemento-osseous dysplasia (COD) based on panoramic radiographs
* Presence of at least one COD-associated tooth suitable for measurement
* Availability of a contralateral healthy tooth to serve as a control
* Teeth with healthy periodontal supporting tissues
* Patients aged ≥18 years
* Patients who have provided written informed consent

Exclusion Criteria:

* Presence of systemic diseases that could affect bone or periodontal structures (e.g., uncontrolled diabetes, osteoporosis, metabolic bone diseases)
* History of radiotherapy or chemotherapy in the head and neck region
* Teeth with extensive caries, mobility, or periodontal disease
* Patients with a history of orthodontic treatment or trauma in the relevant region

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Implant Stability Quotient (ISQ) values by Resonance Frequency Analysis (RFA) | At baseline (single measurement per tooth)
  ISQ values obtained from COD-associated teeth and contralateral healthy teeth using the Osstell™ device. Measurements recorded in mesio-distal and bucco-lingual directions and averaged.

SECONDARY OUTCOMES:
Maximum Bite Force | At baseline (single measurement per tooth)
  Bite force recorded with a bite force sensor to compare functional stability of COD-associated teeth and contralateral healthy teeth.

CONTACTS AND LOCATIONS:
Locations (1):
- Eskişehir Osmangazi University, Eskişehir, Turkey (Türkiye)

REFERENCES:
- [Background] Olive J, Aparicio C. Periotest method as a measure of osseointegrated oral implant stability. Int J Oral Maxillofac Implants. 1990 Winter;5(4):390-400. PMID 2094658
- [Background] Barewal RM, Oates TW, Meredith N, Cochran DL. Resonance frequency measurement of implant stability in vivo on implants with a sandblasted and acid-etched surface. Int J Oral Maxillofac Implants. 2003 Sep-Oct;18(5):641-51. PMID 14579951